CLINICAL TRIAL: NCT01351025
Title: A Pilot Study Evaluating the Effect of Atorvastatin on Biomarkers of Inflammation, Coagulopathy, Angiogenesis, and T-lymphocyte Activation in HIV-1 Infected Individuals With Suppressed HIV-1 RNA and LDL Cholesterol < 130 mg/dL
Brief Title: Atorvastatin on Biomarkers of Inflammation, Coagulopathy, Angiogenesis & T-cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ACTG A5275; 1U01AI068636 (NIH)
Record Dates: First submitted 2010-11-08; First posted 2011-05-10 (Estimated); Results first posted 2015-08-04 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: atorvastatin / placebo (Experimental): At study entry (week 0), participants continued the entry boosted PI-based antiretroviral regimen (not provided by the study) and initiated atorvastatin at a daily dose of 10 mg for 4 weeks. If no symptoms or lab findings suggestive of atorvastatin toxicity were found, the dose of atorvastatin was increased to 20 mg daily at the week 4 visit. At week 20, atorvastatin was stopped for a 4-week washout period.
  At week 24, placebo was started for 4 weeks. If no symptoms or lab findings suggestive of toxicity were found, the placebo dose was doubled at week 28. At week 44, the placebo was stopped to allow for another 4-week washout period.
  Interventions: Drug: atorvastatin; Drug: placebo for atorvastin
- Arm B: placebo / atorvastatin (Experimental): At study entry (week 0), participants continued the entry boosted PI-based antiretroviral regimen (not provided by the study) and initiated placebo for 4 weeks. If no symptoms or lab findings suggestive of toxicity were found, the dose of placebo was doubled at the week 4 visit. At week 20, the placebo was stopped for a 4-week washout period.
  At week 24, atorvastatin was started at a daily dose of 10 mg for 4 weeks. If no symptoms or lab findings suggestive of atorvastatin toxicity were found, the dose of atorvastatin was increased to 20 mg daily at week 28. At week 44, atorvastatin was stopped to allow for another 4-week washout period.
  Interventions: Drug: atorvastatin; Drug: placebo for atorvastin

INTERVENTIONS:
Drug: atorvastatin — 10 mg daily for 4 weeks, if no symptoms or lab findings suggestive of atorvastatin toxicity, dose increase to 20 mg daily from week 4- week 20
  Other Names: Lipitor
  Arms: Arm A: atorvastatin / placebo
Drug: atorvastatin — Starting at week 24, 10 mg daily for 4 weeks. If no symptoms or lab findings suggestive of atorvastatin toxicity were found, 20 mg daily from week 28- week 44.
  Other Names: Lipitor
  Arms: Arm B: placebo / atorvastatin
Drug: placebo for atorvastin — One tablet once daily for 4 weeks. If no symptoms or lab findings suggestive of toxicity were found, then increase the dose to two tablets once daily.
  Other Names: placebo

SUMMARY:
ACTG A5275 was a prospective, double-blind, randomized, placebo-controlled cross-over design pilot study evaluating the effect of atorvastatin on biomarkers of inflammation, coagulopathy, angiogenesis, and T-lymphocyte activation in HIV-1 infected individuals with suppressed HIV-1 RNA on stable protease inhibitor based antiretroviral therapy with fasting LDL cholesterol < 130 mg/dL.

Atorvastatin is a drug approved by the Food and Drug Administration (FDA) for treating high cholesterol. Atorvastatin has also been able to lower the level of inflammation blood tests in certain other diseases but has not been studied for this purpose in people who have HIV. The main goal of this experimental study is to see how taking atorvastatin affects inflammation blood tests in people infected with HIV who do not need to take medicine for high cholesterol. In addition to observing the effects of atorvastatin on the level of inflammation measured in the blood, this study evaluated if atorvastatin is safe for people with HIV who are also taking medication for HIV.

DETAILED DESCRIPTION:
Since people started taking HIV medications, illness from AIDS has decreased, but other serious diseases like heart disease (heart attacks) and certain kinds of cancer have increased. HIV causes inflammation (irritation) inside the body that cannot be felt but can be measured by levels of certain inflammation blood tests. Inflammation may contribute to diseases (such as heart attacks) that have become some of the leading causes of death in people with HIV. HIV therapy can partially lower levels of inflammation measured in blood, however, levels of inflammation in people who have HIV who are taking certain kinds of anti-HIV drugs may remain high compared with those found in people not infected with HIV.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Combination ART that includes any boosted PI regimen for at least 6 months prior to study entry
* No plans to change the antiretroviral regimen in the next year
* Must have been on the same HAART regimen for at least 12 weeks with no change prior to study entry. More information on this criterion can be found in the study protocol.
* If on vitamin D replacement therapy, must have been on stable regimen for ≥ 1 mo. prior to study entry.
* CD4+ T-cell count obtained within 45 days prior to study entry at any laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent.
* Screening HIV-1 RNA < 40 copies/mL by Abbott RealTime PCR at a laboratory certified by the DAIDS Virology Quality Assurance (VQA) program within 45 days prior to study entry.
* All known HIV-1 RNA levels obtained within 180 days prior to study entry are below the limits of quantification on all tests, with documentation of at least 1 test by any FDA-approved assay at a CLIA-certified laboratory obtained between 90 to 180 days prior to study entry. A single RNA "blip" of < 500 copies/mL during this time period was permissible if RNA levels immediately before and after were below the limits of quantification for the assay.
* Laboratory values obtained within 45 days prior to study entry- Absolute neutrophil count (ANC) 750/mm3, Hemoglobin ≥ 9.0 g/dL for female subjects,10.0 g/dL for male subjects, Platelet count ≥ 100,000/mm3, Calculated creatinine clearance (CrCl) 30 mL/min, as estimated by the Cockcroft-Gault equation, Creatine kinase (CK) < 3 x ULN, AST ≤ 2.0 x ULN, ALT ≤ 2.0 x ULN, Total bilirubin ≤ 2.5 x ULN. If the subject was taking an indinavir- or atazanavir-containing regimen at the time of screening, a total bilirubin of ≤ 5 x ULN is acceptable, Fasting LDL cholesterol ≥ 70 mg/dL and < 130 mg/dL, Fasting triglycerides < 400 mg/dL, Fasting glucose < 110 mg/dL
* Screening plasma D-dimer > 0.34 μg/mL from a sample obtained within 45 days prior to study entry was the original D-dimer criterion. It was revised to ≥ 0.25 ug/mL four months after the first enrollment, and subsequently the D-dimer eligibility criterion was completely cut off a year later.
* For females of reproductive potential (women who had not been post-menopausal for at least 24 consecutive months, i.e., who had menses within 24 months prior to study entry), or women who had not undergone surgical sterilization, specifically hysterectomy or bilateral oophorectomy or tubal ligation) required a negative serum or urine pregnancy test within 48 hours prior to entry. More information on this criterion can be found in the study protocol.
* Must agree not to participate in the conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the subject/partner must use at least 2 reliable methods of contraception, (condoms, without a spermicidal agent; a diaphragm or cervical cap without spermicide; an IUD; or hormone-based contraceptive), for 2 weeks before study treatment, while receiving study treatment, and for 6 weeks after receiving study treatment. As hormone-based contraceptives (oral, transdermal, or subdermal) can affect coagulopathy biomarkers, subjects who plan on using such a contraceptive during the study must be taking the same product for ≥ 4 weeks prior to screening and be encouraged to continue throughout the duration of the study if medically feasible.
* Karnofsky performance score ≥ 70 on at least one occasion within 45 days prior to study entry
* Confirmation of the availability of the stored pre-entry fasting plasma, serum, and cell samples. The site had to confirm that these samples had entered into the Laboratory Data Management System (LDMS).

Exclusion Criteria:

* Current or past malignancy (except non-melanoma cancer of the skin)
* Coronary artery disease (CAD) or CAD equivalent including diabetes mellitus or National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) calculated 10-year coronary heart disease (CHD) risk of > 20%.
* Known cirrhosis.
* Known chronic active hepatitis B or C.
* Thyroid-stimulating hormone (TSH) < 1.0 x lower limit of normal or > 1.0 x ULN.
* Known inflammatory conditions, such as, but not limited to, rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), sarcoidosis, inflammatory bowel disease (IBD), chronic pancreatitis, autoimmune hepatitis, myositis, or myopathy.
* Pregnant or breast-feeding.
* Previous intolerance to any statin or any of its components.
* Use of any lipid-lowering therapies including all statin drugs, Omega 3 fatty acids/fish oil, red yeast rice, and niacin products ≥ 1 g/day (e.g., niacin, nicotinic acid, vitamin B3) taken within 45 days prior to study entry. More information on this criterion can be found in the study protocol.
* Immunosuppressant use, such as, but not limited to, systemic or potentially systemic glucocorticoids (including nasal or inhaled steroids), azathioprine, tacrolimus, mycophenolate, sirolimus, rapamycin, or cyclosporine within 45 days prior to study entry.
* Use of any systemic antineoplastic or immunomodulatory treatment, investigational vaccines, interleukins, interferons, growth factors, or intravenous immunoglobulin (IVIG) within 45 days prior to study entry. More information on this criterion can be found in the study protocol.
* Concurrent use of prohibited medications. More information on this criterion can be found in the study protocol.
* Heavy alcohol use as defined by the National Institute on Alcohol Abuse and Alcoholism (NIAAA) (http://pubs.niaaa.nih.gov/publications/Practitioner/pocketguide/pocket_guide3.htm) and alcohol or drug use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Current use of anticoagulation therapy other than ≤ 325 mg of daily aspirin.
* Known coagulopathy, deep venous thrombosis, pulmonary embolism within 6 months prior to study entry.
* Known active or recent (not fully resolved within 4 weeks prior to study entry) bacterial, fungal, parasitic, or viral infections.
* Known history of recurrent rectal and/or genital herpes simplex virus (HSV) or varicella zoster virus (VZV) infection within 12 weeks prior to study entry.
* Serious illness or trauma requiring systemic treatment and/or hospitalization within 4 weeks prior to study entry.
* History of stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-04-14 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A. Aberg, M.D., Study Chair — NYU/Bellevue/HIV/AIDS CTU; Daniel E Nixon, D.O., Ph.D., Study Chair — Virginia Commonwealth University Medical Center
Locations (31):
- United States (30):
  - 31788 Alabama CRS, Birmingham, Alabama
  - UCLA CARE Center CRS (601), Los Angeles, California
  - Ucsd, Avrc Crs (701), San Diego, California
  - Harbor-UCLA Med. Ctr. CRS (603), Torrance, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Georgetown University CRS (GU CRS) (1008), Washington D.C., District of Columbia
  - Northwestern University CRS (2701), Chicago, Illinois
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS (103), Boston, Massachusetts
  - Wayne State Univ. CRS (31478), Detroit, Michigan
  - Henry Ford Hosp. CRS (31472), Detroit, Michigan
  - Washington U CRS (2101), St Louis, Missouri
  - Cooper Univ. Hosp. CRS (31476), Camden, New Jersey
  - New Jersey Medical School-Adult Clinical Research Ctr. CRS (31486), Newark, New Jersey
  - Cornell CRS (7804), New York, New York
  - NY Univ. HIV/AIDS CRS (401), New York, New York
  - AIDS Care CRS (1101), Rochester, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS (31787), Rochester, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS (1601), Durham, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - Metro Health CRS (2503), Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS (2301), Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - Pitt CRS (1001), Pittsburgh, Pennsylvania
  - Houston AIDS Research Team CRS (31473), Houston, Texas
  - Virginia Commonwealth Univ. Medical Ctr. CRS (31475), Richmond, Virginia
  - University of Washington AIDS CRS (1401), Seattle, Washington
- Puerto Rico-AIDS CRS (5401), San Juan, Puerto Rico

REFERENCES:
- [Derived] Rahman F, Brates I, Aweeka F, Bosch RJ, Deitchman A, Nixon D, Aberg JA. Evaluating the effect of atorvastatin exposure and vitamin D levels on lipid outcomes in people with HIV-1 with suppressed HIV-1 RNA and LDL cholesterol <130 mg/dL. HIV Med. 2023 Jun;24(6):749-753. doi: 10.1111/hiv.13453. Epub 2022 Dec 22. PMID 36549898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A5275 opened under version 1.0 on April 7, 2011, and the first participant was randomized on April 14, 2011. Accrual to the study closed on May 31, 2013, with a total of 98 participants enrolled at 31 sites.
Pre-assignment Details: Four enrolled participants did not start study treatment (3 from arm A and 1 from arm B) due to enrollment error and noncompliance. These 4 participants were not included in the study efficacy or safety analyses.
Groups:
- Arm A: Atorvastatin / Placebo: At study entry (week 0), participants continued the entry boosted PI-based antiretroviral regimen (not provided by the study) and initiated atorvastatin at a daily dose of 10 mg for 4 weeks. If no symptoms or lab findings suggestive of atorvastatin toxicity were found, the dose of atorvastatin was increased to 20 mg daily at the week 4 visit. At week 20, atorvastatin was stopped for a 4-week washout period.
  At week 24, placebo was started for 4 weeks. If no symptoms or lab findings suggestive of toxicity were found, the placebo dose was doubled at week 28. At week 44, the placebo was stopped to allow for another 4-week washout period.
  atorvastatin: 10 mg daily for 4 weeks, if no symptoms or lab findings suggestive of atorvastatin toxicity, dose increase to 20 mg daily from week 4 - week 20
- Arm B: Placebo / Atorvastatin: At study entry (week 0), participants continued the entry boosted PI-based antiretroviral regimen (not provided by the study) and initiated placebo for 4 weeks. If no symptoms or lab findings suggestive of toxicity were found, the dose of placebo was doubled at the week 4 visit. At week 20, the placebo was stopped for a 4-week washout period.
  At week 24, atorvastatin was started at a daily dose of 10 mg for 4 weeks. If no symptoms or lab findings suggestive of atorvastatin toxicity were found, the dose of atorvastatin was increased to 20 mg daily at week 28. At week 44, atorvastatin was stopped to allow for another 4-week washout period.
  atorvastatin: Starting at week 24, 10 mg daily for 4 weeks. If no symptoms or lab findings suggestive of atorvastatin toxicity were found, 20 mg daily from week 28- week 44.
Period: Week 0 - 20
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Started | 46 | 48
Completed | 43 | 47
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Week 20 - 24
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Started | 43 | 47
Completed | 43 | 47
Not Completed | 0 | 0
Period: Week 24 - 44
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Started | 43 | 47
Completed | 42 | 43
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Site closed | 0 | 1
Not completed — unable to get to clinic | 1 | 1
Period: Week 44 - 48
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Started | 42 | 43
Completed | 42 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who started study treatment are included
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [39 to 55] | 50 [42 to 55] | 48 [41 to 55]
Age, Customized [Number; unit: participants]
  18-29 Years | 3 | 2 | 5
  30-39 Years | 9 | 6 | 15
  40-49 Years | 16 | 16 | 32
  50-59 Years | 14 | 21 | 35
  >=60 Years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 29 | 35 | 64
Race/Ethnicity, Customized [Number; unit: participants]
  White non-Hispanic | 10 | 13 | 23
  Black non-Hispanic | 21 | 22 | 43
  Hispanic (regardless of race) | 14 | 13 | 27
  Asian, Pacific Islander | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 46 | 48 | 94
HIV-1 RNA [Number; unit: participants]
  < assay lower limit | 46 | 47 | 93
  >= assay lower limit | 0 | 1 | 1
CD4 count [Median (Inter-Quartile Range); unit: cells/mm^3] | 587 [373 to 732] | 545 [424 to 689] | 552 [412 to 714]

OUTCOME MEASURES:

1. Primary Outcome: Difference Between [Change From Week 24 to Week 44] and [Change From Baseline to Week 20] in log10 IL-6
Description: IL-6 (Interleukin 6) in log10 pg/mL: Difference between [change from week 24 to week 44] and [change from baseline to week 20] (i.e. [week 44 - week 24] - [week 20 - baseline])
Time Frame: baseline, week 20, week 24, and week 44
Population: The primary analysis was as-treated, limited to participants who had data for baseline, week 20, week 24, and week 44, and remained on study treatment through week 44 (allowing treatment interruption < 4 weeks), and did not use prohibited medications or have virologic failure during the course of the study.
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Number analyzed (Participants) | 34 | 36
log10 pg/mL | -0.08 [-0.32 to 0.22] | -0.08 [-0.28 to 0.12]
Statistical Analysis 1: Comparison: Arm A: Atorvastatin / Placebo vs Arm B: Placebo / Atorvastatin; The null hypothesis is that there is no difference between arm A and arm B in the differences of the changes ([week 44 - week 24] - [week 20 - baseline]) in log10 IL-6; Test type: Superiority or Other; p = 0.94, Wilcoxon (Mann-Whitney) — Two-sided p-values of < 0.05 without adjustments for multiple testing were considered statistically significant; Exact Wilcoxon rank sum test was used

2. Primary Outcome: Difference Between [Change From Week 24 to Week 44] and [Change From Baseline to Week 20] in CD4+ T-cell Activation Percent
Description: CD4+ T-cell activation percent (% CD38+/DR+ of CD4+): Difference between [change from week 24 to week 44] and [change from baseline to week 20] (i.e. [week 44 - week 24] - [week 20 - baseline])
Time Frame: baseline, week 20, week 24, and week 44
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Number analyzed (Participants) | 31 | 34
percent | -0.20 [-5.00 to 2.20] | 0.60 [-2.90 to 2.40]
Statistical Analysis 1: Comparison: Arm A: Atorvastatin / Placebo vs Arm B: Placebo / Atorvastatin; The null hypothesis is that there is no difference between arm A and arm B in the differences of the changes ([week 44 - week 24] - [week 20 - baseline]) in CD4+ T-cell activation percent (% CD38+/DR+ of CD4); Test type: Superiority or Other; p = 0.495, Wilcoxon (Mann-Whitney) — Two-sided p-values of < 0.05 without adjustments for multiple testing were considered statistically significant; exact Wilcoxon rank sun test was used

3. Primary Outcome: Difference Between [Change From Week 24 to Week 44] and [Change From Baseline to Week 20] in log10 D-dimer
Description: D-dimer in log10 ng/mL: Difference between [change from week 24 to week 44] and [change from baseline to week 20] (i.e. [week 44 - week 24] - [week 20 - baseline])
Time Frame: baseline, week 20, week 24, and week 44
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Number analyzed (Participants) | 34 | 36
log10 ng/mL | -0.02 [-0.13 to 0.14] | 0.00 [-0.18 to 0.08]
Statistical Analysis 1: Comparison: Arm A: Atorvastatin / Placebo vs Arm B: Placebo / Atorvastatin; The null hypothesis is that there is no difference between arm A and arm B in the differences of the changes ([week 44 - week 24] - [week 20 - baseline]) in log10 D-dimer; Test type: Superiority or Other; p = 0.704, Wilcoxon (Mann-Whitney) — Two-sided p-values of < 0.05 without adjustments for multiple testing were considered statistically significant; exact Wilcoxon rank sum test was used

4. Primary Outcome: Difference Between [Change From Week 24 to Week 44] and [Change From Baseline to Week 20] in CD8+ T-cell Activation Percent
Description: CD8+ T-cell activation percent (% CD38+/DR+ of CD8+): Difference between [change from week 24 to week 44] and [change from baseline to week 20] (i.e. [week 44 - week 24] - [week 20 - baseline])
Time Frame: baseline, week 20, week 24, and week 44
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Number analyzed (Participants) | 31 | 34
percent | 1.10 [-4.40 to 5.80] | -1.15 [-4.90 to 3.90]
Statistical Analysis 1: Comparison: Arm A: Atorvastatin / Placebo vs Arm B: Placebo / Atorvastatin; The null hypothesis is that there is no difference between arm A and arm B in the differences of the changes ([week 44 - week 24] - [week 20 - baseline]) in CD8+ T-cell activation percent (% CD38+/DR+ of CD8+); Test type: Superiority or Other; p = 0.508, Wilcoxon (Mann-Whitney) — Two-sided p-values of < 0.05 without adjustments for multiple testing were considered statistically significant; Exact Wilcoxon rank sum test was used

5. Secondary Outcome: Difference Between [Change From Week 24 to Week 44] and Change From [Baseline to Week 20] in MCP-1 (log10 Transformed)
Description: Monocyte chemoattractant protein-1 (MCP-1/CCL2) is one of the key chemokines that regulate migration and infiltration of monocytes/macrophages.
  Difference between [change from week 24 to week 44] and change from [baseline to week 20] is defined as [week 44 - week 24] - [week 20 - baseline].
Time Frame: baseline, week 20, week 24, and week 44
Population: This analysis was as-treated, limited to participants who had data for baseline, week 20, week 24, and week 44, and remained on study treatment through week 44 (allowing treatment interruption < 4 weeks), and did not use prohibited medications or have virologic failure during the course of the study.
Measure: Median (Inter-Quartile Range); unit: log10 pg/ml
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Number analyzed (Participants) | 34 | 36
log10 pg/ml | 0.03 [-0.09 to 0.13] | -0.04 [-0.10 to 0.06]

6. Secondary Outcome: Difference Between [Change From Week 24 to Week 44] and Change From [Baseline to Week 20] in IP-10 (log10 Transformed)
Description: IFN-gamma-inducible protein 10 (IP-10 or CXCL10) is a chemokine secreted from cells stimulated with type I and II IFNs and LPS, is also a chemoattractant for activated T cells.
  Difference between [change from week 24 to week 44] and change from [baseline to week 20] is defined as [week 44 - week 24] - [week 20 - baseline].
Time Frame: baseline, week 20, week 24, and week 44
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: log10 pg/ml
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Number analyzed (Participants) | 34 | 36
log10 pg/ml | -0.03 [-0.10 to 0.14] | -0.04 [-0.09 to 0.06]

7. Secondary Outcome: Difference Between [Change From Week 24 to Week 44] and Change From [Baseline to Week 20] in CD40L (log10 Transformed)
Description: Cluster of differentiation 40 (CD40L) is a costimulatory protein found on antigen presenting cells and is required for their activation.
  Difference between [change from week 24 to week 44] and change from [baseline to week 20] is defined as [week 44 - week 24] - [week 20 - baseline].
Time Frame: baseline, week 20, week 24, and week 44
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: log10 pg/ml
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Number analyzed (Participants) | 34 | 36
log10 pg/ml | 0.01 [-0.18 to 0.20] | -0.03 [-0.17 to 0.08]

8. Secondary Outcome: Difference Between [Change From Week 24 to Week 44] and Change From [Baseline to Week 20] in sCD14 (log10 Transformed)
Description: Soluble cluster of differentiation 14 (sCD14) is a human gene. Difference between [change from week 24 to week 44] and change from [baseline to week 20] is defined as [week 44 - week 24] - [week 20 - baseline].
Time Frame: baseline, week 20, week 24, and week 44
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: log10 ng/ml
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Number analyzed (Participants) | 34 | 36
log10 ng/ml | 0.00 [-0.04 to 0.08] | 0.00 [-0.08 to 0.09]

9. Secondary Outcome: Difference Between [Change From Week 24 to Week 44] and Change From [Baseline to Week 20] in P-selectin (log10 Transformed)
Description: P-selectin is a protein that in humans encoded by the SELP gene. P-selectin functions as a cell adhesion molecule (CAM) on the surfaces of activated endothelial cells, which line the inner surface of blood vessels, and activated platelets.
  Difference between [change from week 24 to week 44] and change from [baseline to week 20] is defined as [week 44 - week 24] - [week 20 - baseline].
Time Frame: baseline, week 20, week 24, and week 44
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: log10 ng/ml
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Number analyzed (Participants) | 34 | 36
log10 ng/ml | 0.01 [-0.10 to 0.17] | -0.06 [-0.14 to 0.05]

10. Secondary Outcome: Difference Between [Change From Week 24 to Week 44] and Change From [Baseline to Week 20] in sCD163 (log10 Transformed)
Description: CD163 (Cluster of Differentiation 163) is a protein that in humans encoded by the CD163 gene; and sCD163 is soluble CD163.
  Difference between [change from week 24 to week 44] and change from [baseline to week 20] is defined as [week 44 - week 24] - [week 20 - baseline].
Time Frame: baseline, week 20, week 24, and week 44
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: log10 ng/ml
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Number analyzed (Participants) | 34 | 36
log10 ng/ml | -0.04 [-0.12 to 0.05] | 0.03 [-0.06 to 0.15]

11. Secondary Outcome: Number of Participants With Safety Endpoints Before Study Treatment Cross-over (Baseline to Week 24)
Description: Safety endpoints are defined as grade ≥ 2 signs and symptoms, laboratory abnormalities, AST/ALT > 3 X ULN, and adverse events prior to study treatment cross-over (baseline to week 24).
  The DAIDS Adverse Event (AE) Grading Table, Version 1.0, December 2004 (Clarification, August 2009) was used for grading of AEs.
Time Frame: week 0 to week 24
Population: participants who started study treatment
Measure: Number; unit: participants
Groups:
- Arm A: Atorvastatin / Placebo: At study entry (week 0), participants continued the entry boosted PI-based antiretroviral regimen (not provided by the study) and initiated atorvastatin at a daily dose of 10 mg for 4 weeks. If no symptoms or lab findings suggestive of atorvastatin toxicity were found, the dose of atorvastatin was increased to 20 mg daily at the week 4 visit. At week 20, atorvastatin was stopped for a 4-week washout period.
  atorvastatin: 10 mg daily for 4 weeks, if no symptoms or lab findings suggestive of atorvastatin toxicity, dose increase to 20 mg daily from week 4 - week 20
- Arm B: Placebo / Atorvastatin: At study entry (week 0), participants continued the entry boosted PI-based antiretroviral regimen (not provided by the study) and initiated placebo for 4 weeks. If no symptoms or lab findings suggestive of toxicity were found, the dose of placebo was doubled at the week 4 visit. At week 20, the placebo was stopped for a 4-week washout period.
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Number analyzed (Participants) | 46 | 48
participants | 20 | 22

12. Secondary Outcome: Number of Participants With Safety Endpoints After Study Treatment Cross-over (Week 24 to Week 48)
Description: Safety endpoints are defined as grade ≥ 2 signs and symptoms, laboratory abnormalities, AST/ALT > 3 X ULN, and adverse events after study treatment cross-over (week 24 to week 48).
  The DAIDS Adverse Event (AE) Grading Table, Version 1.0, December 2004 (Clarification, August 2009) was used for grading of AEs.
Time Frame: week 24 to week 48
Population: participants who crossed over study treatment at week 24
Measure: Number; unit: participants
Groups:
- Arm A: Atorvastatin / Placebo: At week 24, placebo was started for 4 weeks. If no symptoms or lab findings suggestive of toxicity were found, the placebo dose was doubled at week 28. At week 44, the placebo was stopped to allow for another 4-week washout period.
- Arm B: Placebo / Atorvastatin: At week 24, atorvastatin was started at a daily dose of 10 mg for 4 weeks. If no symptoms or lab findings suggestive of atorvastatin toxicity were found, the dose of atorvastatin was increased to 20 mg daily at week 28. At week 44, atorvastatin was stopped to allow for another 4-week washout period.
  atorvastatin: Starting at week 24, 10 mg daily for 4 weeks. If no symptoms or lab findings suggestive of atorvastatin toxicity were found, 20 mg daily from week 28- week 44.
Arm/Group | Arm A: Atorvastatin / Placebo | Arm B: Placebo / Atorvastatin
Number analyzed (Participants) | 41 | 43
participants | 20 | 14

ADVERSE EVENTS:
Time Frame: Week 0 to week 24 (before cross-over) and week 24 to week 48 (after cross-over)
Description: Wk 0-24 and Wk 24-48 summaries included participants started study rx and participants remained on study rx at wk24, respectively. Protocol required reporting of signs/symptoms/lab values of Gr 2+, events led to a change in study rx, and new diagnoses identified by the ACTG criteria. See DAIDS AE Grading Table v.1, Dec04 (Clarification Aug09).
Groups:
- Arm A: Atorvastatin / Placebo Before Cross-over (Week 0 - 24): At study entry (week 0), participants continued the entry boosted PI-based antiretroviral regimen (not provided by the study) and initiated atorvastatin at a daily dose of 10 mg for 4 weeks. If no symptoms or lab findings suggestive of atorvastatin toxicity were found, the dose of atorvastatin was increased to 20 mg daily at the week 4 visit. At week 20, atorvastatin was stopped for a 4-week washout period.
- Arm B: Placebo / Atorvastatin Before Cross-over (Week 0 - 24): At study entry (week 0), participants continued the entry boosted PI-based antiretroviral regimen (not provided by the study) and initiated placebo for 4 weeks. If no symptoms or lab findings suggestive of toxicity were found, the dose of placebo was doubled at the week 4 visit. At week 20, the placebo was stopped for a 4-week washout period.
- Arm A: Atorvastatin / Placebo After Cross-over (Week 24 - 48): At week 24, placebo was started for 4 weeks. If no symptoms or lab findings suggestive of toxicity were found, the placebo dose was doubled at week 28. At week 44, the placebo was stopped to allow for another 4-week washout period.
- Arm B: Placebo / Atorvastatin After Cross-over (Week 24 - 48): At week 24, atorvastatin was started at a daily dose of 10 mg for 4 weeks. If no symptoms or lab findings suggestive of atorvastatin toxicity were found, the dose of atorvastatin was increased to 20 mg daily at week 28. At week 44, atorvastatin was stopped to allow for another 4-week washout period.
Arm/Group | Arm A: Atorvastatin / Placebo Before Cross-over (Week 0 - 24) | Arm B: Placebo / Atorvastatin Before Cross-over (Week 0 - 24) | Arm A: Atorvastatin / Placebo After Cross-over (Week 24 - 48) | Arm B: Placebo / Atorvastatin After Cross-over (Week 24 - 48)
Serious Adverse Events (participants affected / at risk) | 4/46 | 3/48 | 0/41 | 0/43
Other Adverse Events (participants affected / at risk) | 37/46 | 44/48 | 30/41 | 31/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Atorvastatin / Placebo Before Cross-over (Week 0 - 24) (N=46) | Arm B: Placebo / Atorvastatin Before Cross-over (Week 0 - 24) (N=48) | Arm A: Atorvastatin / Placebo After Cross-over (Week 24 - 48) (N=41) | Arm B: Placebo / Atorvastatin After Cross-over (Week 24 - 48) (N=43)
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Atorvastatin / Placebo Before Cross-over (Week 0 - 24) (N=46) | Arm B: Placebo / Atorvastatin Before Cross-over (Week 0 - 24) (N=48) | Arm A: Atorvastatin / Placebo After Cross-over (Week 24 - 48) (N=41) | Arm B: Placebo / Atorvastatin After Cross-over (Week 24 - 48) (N=43)
Fatigue (General disorders) | 2 | 5 | 3 | 0
Alanine aminotransferase abnormal (Investigations) | 1 | 3 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 3 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 1 | 0 | 1
Blood bicarbonate decreased (Investigations) | 1 | 5 | 0 | 1
Blood bilirubin increased (Investigations) | 19 | 24 | 8 | 20
Blood cholesterol increased (Investigations) | 12 | 23 | 15 | 4
Blood creatinine increased (Investigations) | 1 | 8 | 2 | 7
Blood glucose decreased (Investigations) | 4 | 5 | 3 | 2
Blood glucose increased (Investigations) | 3 | 9 | 7 | 6
Blood potassium decreased (Investigations) | 3 | 3 | 3 | 1
Low density lipoprotein increased (Investigations) | 7 | 18 | 8 | 0
Platelet count decreased (Investigations) | 3 | 2 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 4
Headache (Nervous system disorders) | 4 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.